CLINICAL TRIAL: NCT03421951
Title: A Prospective Single-arm, Multi-center Clinical Study Examining the Changes in Quality of Life and Pain Following Dorsal Root Ganglion Stimulation for the Treatment of Chronic Intractable Pelvic and Lower Limb Pain
Brief Title: Change in Pain and Quality of Life Following SCS for Chronic Pain
Acronym: BURST
Status: Terminated | Type: Observational
Why Stopped: Sponsor withdrew funding
Sponsor: KM Clinical Research Group (Industry)
Responsible Party: Principal Investigator, Kate McLellan, Principle Investigator, KM Clinical Research Group
Other Study IDs: 2017-PN-02
Record Dates: First submitted 2018-01-30; First posted 2018-02-05 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Pain, Chronic; Pain, Radiating; Pain, Back; Pain Syndrome
Keywords: spine; lower limb
MeSH Terms: conditions — Chronic Pain; Pain; Back Pain; Somatoform Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study Title Subject-reported treatment efficacy and procedure satisfaction (steps) study.BURST study- a prospective observational clinical study examining the changes in quality of life and pain following spinal cord stimulation for the treatment of chronic intractable lower back and lower limb pain.

DETAILED DESCRIPTION:
Objectives The primary objective is changes in lower back and/or lower limb pain patient-reported satisfaction with procedure outcome and treatment efficacy to reduce pain levels following an orthopedic procedure for knees, hips, shoulders, elbows, wrists, or anklesspinal cord (SCS) stimulation. Secondary objectives include changes in physical health, quality of life, and quality of life and pain-related prescription medication usage.

Design and Outcomes This is a prospective observational single-arm study to access the primary outcome variable of lower back and/or lower limb patient satisfaction with procedure outcomes as measured using a modified MacNab scale. Patients will have presented to their healthcare providers with knee, hip, shoulder, elbow, wrist, or ankle pain and will have elected and been assigned a medically-appropriate surgical procedure as part of their standard of care. It is possible for subjects to have multiple areas of pain and subsequent surgeries, and subjects have the option of completing surveys for all medically-indicatedmedically indicated areas being treated.pain

IIIntervention and Duration There will be no study intervention. Subjects will only be monitored and evaluated for pre and post-operative satisfaction, pain, physical activity levels, quality of life, and medication use levels. Subjects will be followed for 12 months following their SCS stimulation implant procedure.

Sample Size and Population Investigators aim for a minimum population size of 1,500 in order to give statistical significance with results. Subjects will be stratified by surgical procedurearea of chronic pain.

ELIGIBILITY:
Inclusion Criteria:

Prescribed spinal cord stimulator implant by their healthcare provider. Previous conservative care such as physical therapy or chiropractic care that failed to provide adequate pain relief.

Willing and able to adhere to the protocol of the study including the survey timeline.

Between the ages of 18-85 years.

Exclusion Criteria:

Unwilling to sign Informed Consent and comply with protocol

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will be patients who have already been prescribed a trial spinal cord stimulator implant procedure to treat their lower back or lower limb pain.
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Change in Pain Levels | 12 months post-permanent spinal cord stimulator implantation
  Change in self-reported pain levels
Change in quality of life | 12 months post-permanent spinal cord stimulator implantation
  change in self-reported quality of life

SECONDARY OUTCOMES:
Change in prescription pain medication use | 12 months post-permanent spinal cord stimulator implantation
  change in opioid medication use to control pain

CONTACTS AND LOCATIONS:
Overall Officials: Kate McLellan, PhD, Study Director — KM Clinical Research Group
Locations (1):
- KM Clinical Research Group, Murrieta, California, United States